CLINICAL TRIAL: NCT02172716
Title: Disruption of Immune Homeostasis in Type 2 Diabetics With Generalized Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Augusta University (Other)
Responsible Party: Principal Investigator, Giuseppe Alexandre Romito, Professor and Chair, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26793214.9.0000.0075
Record Dates: First submitted 2014-06-17; First posted 2014-06-24 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 2; Type 2 Diabetes Mellitus; Periodontal Diseases; Periodontitis; Chronic Periodontitis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Periodontal Diseases; Periodontitis; Chronic Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nonsurgical periodontal treatment (Experimental): Nonsurgical periodontal treatment will be conducted following a full-mouth approach; no antibiotics or chemical plaque control will be provided.
  Interventions: Procedure: Nonsurgical periodontal treatment

INTERVENTIONS:
Procedure: Nonsurgical periodontal treatment — All patients with GCP will receive full-mouth scaling and root planning under local analgesia in one session. Hopeless teeth will be treated similarly and extracted after de 30 days visit. Oral hygiene instructions will be given as needed.
  Supragingival scaling Periodontally healthy subjects will receive supra-gingival scaling and polishing in one appointment as needed. Oral hygiene instructions will be given as needed.

SUMMARY:
The primary objective of this study is to assess the short-term immune response of type-2 diabetics with generalized chronic periodontitis (GCP) to nonsurgical periodontal treatment.

The investigators hypothesize that type-2 diabetes exacerbates the disruption of DC (dendritic cells)-mediated immune homeostasis associated with periodontitis.

DETAILED DESCRIPTION:
Objectives: The primary objective of this study is to assess the short-term immune response of type-2 diabetics with generalized chronic periodontitis (GCP) to nonsurgical periodontal treatment.

Hypothesis: we hypothesize that type-2 diabetes exacerbates the disruption of DC-mediated immune homeostasis associated with periodontitis.

Subject population: Four groups comprising 80 subjects will be selected to participate: type 2 diabetics with GCP (n=20), prediabetics with GCP (n=20), normoglycemics with GCP (n=20) and healthy controls (n=20).

Study design: discovery study nested within a single-arm, single blinded clinical trial.

Experimental periods: Screening/Baseline Visit, Treatment Visit, 24 hours, 30 days and 3 months after treatment.

Intervention: Nonsurgical periodontal treatment will be conducted following a full-mouth approach; no antibiotics or chemical plaque control will be provided.

Primary outcomes:

* Cellular measures: Blood PBMCs- counts of myeloid DC (BDCA-1+CD19-), Plasmacytoid DC (cd123+cd303+) NK (CD56+CD16+), Th17, Treg (CD25+, CD39,CD73,CD127, cd152)
* Molecular measures: (Serum/crevicular fluid/ saliva): Anti-mfa-1 IgG (ELISA), Levels of IDO-1, TGFβ, TNFα, IL-1β, IL-6, IL-2, IL-10, IL-17, IL-23, IFNγ, CXCL12 (SDF1) by Multiplexing Luminex immunoassay [MAGPIX®]), performed in triplicate
* Expression on mDCs by custom qrt-PCR array (One step-fast cycle Taqman®, life technologiesTM of: angiopoietin-2, follistatin, GM-CSF, G-CSF, HGF, IL8, IL-6, leptin, PDGF-BB, PECAM-1, VEGF, TGFβ, IDO-1, IL-10, IL-1β, caspase-1, IL-17, IL-23, IL-23R IL-33, IL-12 p70, TRAIL, FOX01, Bcl-2, CXCL12 (SDF-1), CCL19, CCL21 analyzed in triplicate.
* Secondary outcomes: periodontal probing depth, periodontal attachment level, bleeding on probing, visible plaque and gingival bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 35 and 65 years
2. Subject diagnosed with T2DM (HbA1C ≥6.5), prediabetic (HbA1C ≥5.7 and ≤6.4) and non-diabetic (HbA1C ≤5.6) according to American Diabetes Association, 2013.
3. Subjects with GCP (PPD ≥5 mm in ≥10 teeth and BOP in ≥30% of sites) and without GCP (PPD ≤4mm and BOP in <30% sites)
4. Non-smokers or former smokers ≥5 years after quitting

Exclusion Criteria:

1. Pregnant or lactating women
2. Subjects taking medications known to affect the periodontium including phenytoin, cyclosporine
3. Subjects with immunosuppressive conditions or diseases including HIV infection or Hepatitis (B, C).
4. Subjects who require antibiotic prophylaxis for dental procedures.
5. Subjects who have taken antibiotics in the last 6 months
6. Subjects taking daily NSAIDS or on steroidal anti- inflammatory medications

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cellular measures | 24 hours, 30 days and 3 months after treatment.
  Cellular measures: Blood PBMCs- counts of myeloid DC (BDCA-1+CD19-), Plasmacytoid DC (cd123+cd303+) NK (CD56+CD16+), Th17, Treg (CD25+, CD39,CD73,CD127, cd152)
Change from baseline in molecular measures | 24 hours, 30 days and 3 months after treatment.
  Molecular measures: (Serum/crevicular fluid/ saliva): Anti-mfa-1 IgG (ELISA), Levels of IDO-1, TGFβ, TNFα, IL-1β, IL-6, IL-2, IL-10, IL-17, IL-23, IFNγ, CXCL12 (SDF1) by Multiplexing Luminex immunoassay [MAGPIX®]), performed in triplicate
Change from baseline in the expression on mDCs | 24 hours, 30 days and 3 months after treatment.
  Expression on mDCs by custom qrt-PCR array (One step-fast cycle Taqman®, life technologiesTM of: angiopoietin-2, follistatin, GM-CSF, G-CSF, HGF, IL8, IL-6, leptin, PDGF-BB, PECAM-1, VEGF, TGFβ, IDO-1, IL-10, IL-1β, caspase-1, IL-17, IL-23, IL-23R IL-33, IL-12 p70, TRAIL, FOX01, Bcl-2, CXCL12 (SDF-1), CCL19, CCL21 analyzed in triplicate.

SECONDARY OUTCOMES:
periodontal probing depth, periodontal attachment level, bleeding on probing, visible plaque and gingival bleeding. | Baseline, 30 days and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Romito, PhD, Principal Investigator — Professor and chair; Mariana Rabelo, MSc, Study Chair — Post graduate student
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil